CLINICAL TRIAL: NCT05600439
Title: CareME - Efficacy of an Attachment-based Intervention in Residential Care: A Randomized Controlled Trial on the Effects on the Caregivers' Relational Skills and the Adolescents' Psychosocial Adaptation
Brief Title: Efficacy of an Attachment-based Intervention in Residential Care (CareME)
Acronym: CareME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CareME
Record Dates: First submitted 2022-09-30; First posted 2022-10-31 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Professional Role
Keywords: Attachment, Caregiving, Professionals, Youth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental GP (Experimental): CareME Program. Group attachment-based intervention program developed for improving relational abilities in professional caregivers working in Youth Residential Care (YRC) settings.
  Interventions: Behavioral: CareME
- Control GP (No Intervention): The control group had no intervention assigned.

INTERVENTIONS:
Behavioral: CareME — CareME program was planned to integrate 12 group session (90 minutes), implemented fortnightly during a 6-month period, and facilitated by two psychologists and expert researchers on attachment framework. Components included psychoeducation (description of core concepts such as attachment, secure base, safe haven, emotion regulation, mentalization, trauma, and discussion of research on professional caregiving in YRC); experiential and relational exercises (roleplay; cases discussion, film script discussion).
  The program has 7 moduli: (i) adolescents' "pain-based behaviors" and attachment theoretical lens; (ii) adolescence and main developmental challenges (iii) setting rules and limits; (iv) trust & secure base (figures and environment); (v) professionals' stories of attachment & caregiving (vi) personal and structural characteristics that prevent a secure caregiving environment and (vii) professional impairment and strategies promoting healthy secure base provision.
  Arms: Experimental GP

SUMMARY:
CareME is a group attachment-based intervention program developed for improving relational abilities in professional caregivers working in Youth Residential Care (YRC) settings. The intervention program was planned to integrate 12 group session (90 minutes each), implemented fortnightly during a 6-month period, and facilitated by two psychologists and expertise researchers on attachment framework.

The project aims to produce effects on professional caregivers' behaviors and, as an indirect effect, to produce changes on adolescents' outcomes (age 12 to 18 years old).

Regarding professional caregivers' behaviors the project aims to improve reflective functioning, perspective taking, emotion regulation, group intervention practices and quality of relationships in RC (primary outcomes). Additionally, it's expected to reduce levels of professional exhaustion and improve mental health (secondary outcomes). Attachment was considered a moderator. As a result of professional's caregivers behavior change, it is expected to observe subsequent effects on adolescents' psychosocial adaptation indicators, such as improvements on the quality of relationship with professional caregivers, hope, self-efficacy and in emotional regulations processes and a decrease on antisocial behavior, anger control problems and emotional suffering (secondary outcomes). Attachment was considered also a moderator.

Program efficacy was evaluated using a randomized control trial (RCT). Institutions were assigned to the experimental (n = 10) and to the control (n = 11) group using a covariate adaptative randomization method. Data was assessed using a 4-wave longitudinal design (baseline, interim, post, 6-month follow-up) with professional caregivers and adolescents' self-reports.

DETAILED DESCRIPTION:
CareME is a group attachment-based intervention program developed for improving relational abilities in professional caregivers working in Youth Residential Care (YRC) settings. The intervention program was planned to integrate 12 group session (90 minutes each), implemented fortnightly during a 6-month period, and facilitated by two psychologists and expertise researchers on attachment framework.

Aim CareME highlights the role of relational dynamics with significant figures from the residential care context - the caregivers - as enablers of resilient processes and the adaptive development of young people in face of adversity trajectories. More specifically CareME intends to improve the quality of care provided by professional caregivers, by enhancing relational skills directly associated with sensitive care such as emotional regulation and mentalization and improve caregiving behaviors such as emotional support and autonomy granting. It is also expected that changes on professional relational abilities would have a subsequent effect on adolescents' behavioral problems and socioemotional adaptation dimensions.

The elaboration of the intervention was clearly theoretically grounded, based on J. Bowlby and M. Ainsworth's attachment theory, focusing on the development of secure relationships as protective factors against risk. In this sense, the intervention is framed on the crucial role that these professionals have on providing the emotional secure environment for adolescent's psychosocial adaptation and development, minimizing risk and preventing psychopathology. As in other attachment-based intervention programs relational processes intrinsically associated with attachment dimensions, emotional regulation and mentalization were particularly intentionalized during intervention.

More specifically, the project aims to produce effects on professional caregivers' behaviors and, as an indirect effect, to produce changes on adolescents' outcomes (age 12 to 18 years old). Regarding professional caregivers' behaviors, the project aims to improve reflective functioning, perspective taking, emotion regulation, group intervention practices and quality of relationships in RC. Additionally, it's expected to reduce levels of professional exhaustion, improve mental health. Attachment was considered a moderator. As a result of a professional's caregiver's behavior change, it is expected to observe indirect effects on adolescents' psychosocial adaptation indicators, such as improvements in the quality of relationship with professional caregivers, hope, and self-efficacy and in emotional regulations processes and a decrease on antisocial behavior, anger control problems and emotional suffering (secondary outcomes). Attachment was considered also a moderator.

The intervention was programmed to be conducted in person in the Faculty of Psychology and Sciences of Education from the University of Porto facilities. Nevertheless, there were important changes that were introduced to what was initially programmed. The program periodicity, duration, and number of sessions, were changed due to unpredicted challenges introduced by the 1st wave of the pandemic (March 2020). The first 3 sessions (February/March 2020) were conducted fortnightly in person as planned. Then, there was a 7-month period of interruption due to the abrupt changes introduced by the pandemic. The program restarted in October 2020 online on a weekly basis (7 sessions) ending in December 2020. The interruption period resulted from the implications of lockdown measures on YRC organization, and the need to respond to most pressing needs regarding management (e.g., prevent youth and staff contamination, ensure continued responses to other healthcare and psychological intervention needs, ensure communication between youth and most significative ones as family/other relatives/friends, and ensure conditions for distance education). All sessions were then discussed and evaluated according to the project intervention plan and attachment framework. Sessions were supervised by two expert researchers on psychological intervention implementation.

The project was approved by the Ethical Committee of the Faculty of Psychology and Sciences of Education from the University of Porto and the University of Trás-os-Montes and Alto Douro, Portugal.

Procedure: The project was presented to all YRC managers (directors) from Porto district and a total of 21 from the 24 juvenile residential care facilities from Porto district agreed to participate. The dissemination process was facilitated by the National Social Protection sector from Porto District.

Considering the great variation in YRC facilities assigned to the study, randomization was conducted using a covariate adaptative randomization method. YRC facilities were distributed by the experimental (n = 10) and control (n =11) groups according to the minimization method balancing allocation by house facilities (homes vs institution), house typology (gender-specific and mixed), child to caregiver ratio and a number of caregivers. The sample included a total of 212 professional caregivers aiming to integrate the CareME intervention project (Experimental group = 110 professionals) and Control group = 106). A total of 5 groups were created (n < 25 individuals), integrating elements from multiple YRC from the experimental group. Considering that in most institutions' professional caregivers from the technical staff group have management and hierarchical positions towards the educative group, people were also assigned to each group considering the professional role they have in the institution (technical or educative group).

Data Collection was conducted using a 4-wave longitudinal design (baseline - T0, interim -T1 (seven months), post -T2 (13 months) and follow-up-T3 (19 months), using professional caregivers and adolescents' self-reports. Initially, all data collection was planned to be conducted in person in YRC facilities with the supervision and support from 2 researchers. Due to the pandemic, only the 1st wave/baseline was conducted presential. The first wave (baseline) was conducted from November 2019 to January 2020; the 2nd wave (interim), was conducted from June to September 2020, mainly for capturing/controlling the effects of the pandemic; the 3rd wave was conducted between December 2020 and March 2021. The 4th wave (6-month follow-up) was conducted between July and October 2021.

The general objectives of the study were presented in each administration and standardized instructions were given regarding the assessment procedure. After their written informed consent/assent, data collection was conducted. Participation was voluntary and anonymous, and no financial compensation was involved. During the first wave/baseline, two researchers were available to support data collection and ensure confidentiality/anonymity. Afterward, when necessary, online support was given for supporting data collection.

The control group didn´t have any additional intervention assigned.

ELIGIBILITY:
Inclusion Criteria:

* Professionals from the educative and technical team working in YRC settings from the selected facilities
* Professionals that work with children age ranging 12 and 18 years old.

Exclusion Criteria:

- RC facilities that didn´t sign up at least 70% of professional caregivers (both from the technical and educative team)

For adolescents:

Inclusion Criteria:

* Adolescents currently in YRC facilities
* Adolescents with ages ranging between 12 and 18 years old at the 1st data collection.

Exclusion Criteria:

- Adolescents with severe cognitive or emotional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Reflexive functioning (Professionals) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the Reflective Functioning Questionnaire (RFQ, Fonagy et al., 2016; Neto et al, xxx), for assessing certainty (4 items, e.g., "I don't always know why I do what I do") and uncertainty (4 items, e.g., "I always know what I feel.") regarding self and other mental states. Items are rated using 7-point Likert scale from 1 ("Strongly disagree") to 4 ("Strongly agree") .
Change from Baseline Perspective Taking (Professionals) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the perspective taking scale from Interpersonal Reactivity Index (IRI; Davis, 1980, 1983; Limpo et al., 2010). It consists of 7 items (e.g., Sometimes I have a hard time seeing things from the young people's point of view), rated on 5-point Likert-scale from 1 (does not describe me at all) to 5 (describes me very well).
Change from Baseline Group intervention practices (Professionals) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in Group Care Worker Intervention Checklist - GICL (Bastiaanssen et al., 2012; Santos et al., 2019) for assessing support (6 items, e.g., "Offering individual attention") autonomy (7 items, e.g., "Promote social independence") and control (8 items, e.g., "Learning to obey") rated on 3-point Likert scale from 1 ("not true") to 3 ("true").
Change from Baseline Quality of relationships with YRC (Professionals) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Quality of relationships with YRC (Mota & Matos, 2010 adapted) was used for assessing "Caregiver as a Support figure" (6 items, e.g., "I feel youngsters trust me") and "Fear of merging boundaries" (9 items, e.g., "I feel I give more that I should") rated on a 6 point Likert scale from 1 ("I completely disagree") to 6 ("I completely agree").
Change from Baseline Emotion Regulation (Professionals) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the Affect Regulation Checklist (ARC; Moretti, 2003; Santos et al, submitted). ARC is a 12 items questionnaire that evaluates 3 dimensions: suppression (4 items, e.g., "I try hard not to think about my feelings"), dysregulation (4 items, "My feelings just take over me and I can't do anything about it"), and adaptive reflection (4 items, "Thinking about why I have different feelings helps me to learn about myself"). Items are rated in a 5-point Likert scale ranging from 1 ("Not like me") to 5 ("A lot like me").

SECONDARY OUTCOMES:
Change from Baseline Exhaustion (Professionals)at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the exhaustion scale from the questionnaire Oldenburg Burnout Inventory OLBI (Demerouti & Bakker, 1999; Sinval et al., 2019). It is composed by 8 items (e.g., "There are days when I feel tired before I arrive at work") scored on a 6-point Likert scale ranging from 1 ("I strongly disagree "to 6 ("I strongly agree").
Change from Baseline Mental health (Professionals) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the well-being (4 items; e.g., "I have felt OK about myself"), Symptoms (12 items, e.g.," I have felt tense, anxious or nervous") and Functioning scales (12 items, e.g., "I have been happy with the things I have done") from the Clinical Outcome Routine Evaluation - no risk (CORE-NR; Sales et al., 2012), rated on a 5-point Likert scale from 1("never") to 5 ("always or almost always").
Change from Baseline Quality of relationship with Professional Caregivers (Adolescents)at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the professional caregiver's subscale from Connection Questionnaire to Staff and Teachers (QLFP) - (Mota & Matos, 2005). This subscale aggregates 14 items (14 items, e.g., I feel close to some careworkers of the residential care setting I live in), rated on a 6-point Likert-Scale, from (1) "Strongly Disagree" through (6) "Strongly Agree".
Change from Baseline Hope (Adolescents) at T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the hope scale from Vision About Future (Ginevra et al., 2017; Nunes, et al., 2018). It consists of 10 items (e.g., I feel that I will get along quite well.), rated on 5-point Likert-scale from 1 (does not describe me at all) to 5 (describes me very well).
Change from Baseline Psychological adjustment problems (Adolescents) at T1 (seven months), T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the Reynolds Adolescent Adjustment Screening Inventory (RAASI, Reynolds, 2001, Calheiros et al., 2009). RAASI is 32 items scale that evaluates 4 dimensions Antisocial Behavior (5 items, e.g., "I did things that were against the law"), Anger control problems (11 items "I felt angry"), Emotional distress (10 items e.g., "I worried a lot about the future"), and Positive self (6 items e.g., "I felt good about myself") rated on a 3-point Likert scale, from 1 (never or almost never) to 3 (always or almost always).
Change from Baseline Self-efficacy (Adolescents) at T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the General Self-Efficacy Scale (GSE, Jerusalem & Schwarzer, 1981; Araújo & Moura, 2011). GSE is a 10-item scale that evaluates self-efficacy (e.g., I can always manage to solve difficult if I try hard enough"). Rated on a 4-point Likert scale, from 1 (not all true) to 3 (exactly true).
Change from Baseline Emotion regulation (Adolescents) at T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the scales "do not hide emotions" (e.g., When I am angry or upset' I try to hide this) and "differentiating emotions" (e.g., When I am upset' I don´t know if I am sad' scared or angry) the Emotion Awareness Questionnaire (EAQ) (Rieffe et al., 2007; Veiga, et al., 2017), rated on a 3 point Likert scale from 1 (Not true) to 3 (True).
Change from Baseline Satisfaction with residential setting (Adolescents) at T2 (13 months) and T3 (follow up - 19 months) | baseline
  Participants filled in the Caregiving Environment Satisfaction Questionnaire (McDowall, 2013, adapted by Santos et al., 2019). The scale is composed by 7 items (e.g., "I have the privacy I need") rated on a 4-point Likert scale, from (1) Strongly Disagree to (4) Strongly Agree.
Change from Baseline Attachment (Adolescents) at T1 (seven months) and T2 (13 months) | baseline
  Participants filled in the Vulnerable Attachment Style Questionnaire (VASQ) (Bifulco, et al. 2003, Santos et al., 2019). VASQ is a 22-item scale that evaluates Insecurity (12 items, e.g., It's best not to get too emotionally close to other people) and Proximity-Seeking (10 items, e.g., I rely on others to help me make decisions), rated on a 5-point Likert Scale, from (1) "Strongly Disagree" through (5) "Strongly Agree".

OTHER OUTCOMES:
Change from Baseline Attachment (Professionals) at T3 (follow up - 19 months) | baseline
  Participants filled in the Experiences in Close Relationships - Relationship Structures Questionnaire (ECR-RS, Fraley et al., 2011; Moreira et al., 2015). ECR is 9 item scale composed by attachment-related anxiety (3 items, e.g., "I worry that romantic partners won't care about me as much as I care about them") and avoidance (6 items, e.g., "I prefer not to show a partner how I feel deep down"). Each item was scored on a 7-point Likert scale ranging from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina P Mota, PhD, Principal Investigator — University of Trás-os-Montes and Alto Douro
Locations (1):
- University of Trás-os-Montes and Alto Douro, Vila Real, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After project completion.
Access Criteria: Use for research purposes.

REFERENCES:
- [Background] Ainsworth, M. S., & Bowlby, J. (1991). An ethological approach to personality development. American psychologist, 46(4), 333.
- [Background] Bowlby, J. (1973). Attachment and loss: Volume II: Separation, anxiety and anger. In Attachment and loss: Volume II: Separation, anxiety and anger (pp. 1-429). The Hogarth press and the institute of psycho-analysis.
- [Background] Bowlby, J. (1988). A secure base: Parent-child attachment and healthy human development. Basic Books.
- [Background] Fonagy, P., Gergely, G., Jurist, E. L., & Target, M. (2018). Affect regulation, mentalization, and the development of the self. Routledge.
- [Background] Moretti MM, Obsuth I, Craig SG, Bartolo T. An attachment-based intervention for parents of adolescents at risk: mechanisms of change. Attach Hum Dev. 2015;17(2):119-35. doi: 10.1080/14616734.2015.1006383. Epub 2015 Mar 18. PMID 25782460
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Törrönen, M. (2021). Social relationships and their connection to mental health for young people who have been in the care system. The British Journal of Social Work, 51. https://doi.org/10.1093/bjsw/bcab028
- [Background] Zegers MA, Schuengel C, Van IJzendoorn MH, Janssens JM. Attachment and problem behavior of adolescents during residential treatment. Attach Hum Dev. 2008 Mar;10(1):91-103. doi: 10.1080/14616730701868621. PMID 18351496
- [Result] Costa M, Matos PM, Santos B, Carvalho H, Ferreira T, Mota CP. We stick together! COVID-19 and psychological adjustment in youth residential care. Child Abuse Negl. 2022 Aug;130(Pt 1):105370. doi: 10.1016/j.chiabu.2021.105370. Epub 2021 Oct 18. PMID 34756741
- See also: CareME outputs — https://zenodo.org/communities/careme/?page=1&size=20